CLINICAL TRIAL: NCT04680325
Title: Impact of Cranberry Juice Consumption on Gut and Vaginal Microbiota in Post-menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas, Fayetteville (Other)
Collaborators: Ocean Spray, Inc. (Industry)
Responsible Party: Principal Investigator, Franck, Assistant Professor, University of Arkansas, Fayetteville
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Ocean Spray
Record Dates: First submitted 2020-12-16; First posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo juice (Placebo Comparator)
  Interventions: Dietary Supplement: Juice daily consumption
- Cranberry juice (Active Comparator)
  Interventions: Dietary Supplement: Juice daily consumption

INTERVENTIONS:
Dietary Supplement: Juice daily consumption — Single-service bottles of juice were provided for 15 days of daily consumption in each arm

SUMMARY:
This study was a randomized, placebo-controlled, crossover, pilot dietary intervention. Ocean Spray Cranberries, Inc provided the experimental and placebo beverages, which have been validated and used in previous studies [26-29]. Both beverages were similar in appearance, taste, and aroma and assigned to volunteers according to computer-generated random orders. Both investigators and participants were blind to the assignment and products are identified by a random 3-digit code pre-printed on the cap. The participants consumed either cranberry juice or placebo beverage daily (8 fl oz per day) for 15 days

DETAILED DESCRIPTION:
This was a prospective exploratory pilot study with a dietary intervention. Twenty-three (23) women volunteered and participated in this study. The eligibility (no menstrual period for at least 12 months) of the participants was determined using a questionnaire. The participants were postmenopausal women between the ages of 50-75 years old who met the exclusion criteria including no recent antibiotics or immunosuppressive therapies, surgery of the stomach, small or large intestines, appendectomy, gastric bypass or gastric banding in the previous 6 months, and diagnostic with any autoimmune diseases.

This study was a randomized, placebo-controlled, crossover, pilot dietary intervention. Ocean Spray Cranberries, Inc provided the experimental and placebo beverages, which have been validated and used in previous studies [26-29]. Both beverages were similar in appearance, taste, and aroma and assigned to volunteers according to computer-generated random orders. Both investigators and participants were blind to the assignment and products are identified by a random 3-digit code pre-printed on the cap. The participants consumed either cranberry juice or placebo beverage daily (8 fl oz per day) for 15 days

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal status

Exclusion Criteria:

* recent (6months) antibiotics or immunosuppressive therapies
* recent (6months) abdominal surgeries

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Based on menopausal status
Enrollment: 23 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Changes in the vaginal microbiota profile assessed by sequencing of swab samples | 4 weeks
Changes in the gut microbiota profile assessed by sequencing of stool samples | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Franck Carbonero, Principal Investigator — Washington State University
Locations (1):
- University of Arkansas, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No